CLINICAL TRIAL: NCT03015155
Title: Effect of Local Myocardial Hypothermia on Outcomes in Patients With Acute Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention.
Brief Title: Therapeutic Effect of Local Hypothermia in Treatment of Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LS-81570363
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-12

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia (Experimental): Infusion of Cold Saline into Local Infarction Myocardium. A standard working guide-wire, Runthrough NS (Terumo, Japan), is advanced into the distal part of the target coronary artery by using angiography. Compared to the standard PPCI after the balloon expansion, the aspirated catheter (Diver C.E. MAX, Italy) is firstly placed at the location of the distal occlusion lesion to achieve local myocardial hypothermia by infusing the cold saline (4℃, 2.5ml/min, 5min). Then we retract the aspirated catheter, following the balloon expansion and the drug eluting stent implanting. Subsequently, the infusion catheter is tautologically placed at the location of the opened occlusion, within the stent, to persistently perfuse the infarct myocardium with cold saline (4℃, 2.5ml/min, 15min).
  Interventions: Procedure: Infusion of Cold Saline into Local Infarction Myocardium.
- Standard treatment (No Intervention): We place a standard working guide-wire, Runthrough NS (Terumo Corporation, Japan), crossover the criminal lesion of to the distal of the target coronary artery after angiography. Then the pre-dilated balloon is placed at the occluded lesion site to expand the criminal vessel without hypothermia intervention. The operation will be completed when the flow of target coronary artery achieves TIMI class 3 after the drug eluting stent implanting.

INTERVENTIONS:
Procedure: Infusion of Cold Saline into Local Infarction Myocardium. — Infusion of Cold Saline into the Area of Ischemic Myocardium by Using Aspirated Catheter Before the Ischemia/reperfusion.
  Arms: Hypothermia

SUMMARY:
Recent clinical studies have shown that systemic therapeutic hypothermia improving the outcomes in patients with ST segment elevated myocardial infarction (STEMI) received primary percutaneous coronary intervention (P-PCI).Likewise, a few in vivo animal experiments have described the methods, mechanism and rationale of therapeutic hypothermia, including local myocardial hypothermia. However, little is known of the local myocardial hypothermia having impact on prognosis of the patients with acute myocardial infarction. The aim of this study is to ascertain whether local myocardial hypothermia is effective in treatment of ischemia/reperfusion injury in patients with STEMI undergoing P-PCI.

DETAILED DESCRIPTION:
Ethics and organization The study was designed in agreement with the Declaration of Nanjing, and the study protocol was approved by the local ethics committees. A written informed consent will be completed before inclusion. The trial was coordinated and monitored by the First Affiliated Hospital with Nanjing Medical University. An independent data and safety monitoring board, including of physicians independent of the trial sponsor and operational leadership, monitored the safety of the study.

Study population From March 2017 to March 2019, 300 patients from department of cardiology (the First Affiliated Hospital with Nanjing Medical University, Nanjing, China) will be enrolled in this prospective, randomized, end point-blinded study to evaluate the local hypothermia as an adjunct therapy in patients with acute myocardial infarction (AMI) eligible for primary percutaneous intervention (PPCI). Men and women ages 40 and 80 years presenting with anterior or non-anterior AMIs with ST-segment elevation>0.2 mV in 2 contiguous leads and a duration of symptoms<12h will be included. We will collect a second electrocardiogram in the catheterization laboratory before randomization to ensure persistent ST-segment elevation. We conduct the exclusive criterion, including patients with previous AMIs, previous PCI or coronary artery bypass grafting, congestive heart failure, end-stage kidney disease or hepatic failure, recent stroke, coagulopathy, pregnancy, cardiac arrest, or Killip class II to IV at presentation.

Protocol. The AMI patients will be randomized 1:1 to hypothermia or standard of care before coronary angiography. Using varying block sizes and stratification, we generate the randomization list by computer. A standard working guide-wire, Runthrough NS (Terumo Corporation, Japan), is advanced into the distal part of the target coronary artery after determining of the criminal vessel by using angiography. Compared to the standard PPCI after the balloon expansion, the aspirated catheter (Diver C.E. MAX, Invatec S.p.A, Italy) is firstly placed at the location of the distal occlusion lesion to achieve local myocardial hypothermia by infusing the cold saline (4℃, 2.5ml/min, 5min). Then we retract the aspirated catheter, following the balloon expansion and the drug eluting stent implanting. Subsequently, the infusion catheter is tautologically placed at the location of the opened occlusion, within the stent, to persistently perfuse the infarct myocardium with cold saline (4℃, 2.5ml/min, 15min). Loading doses of 300 mg of aspirin, 180 mg ticagrelor and heparin (100u/kg) will be given to all patients before cardiac catheterization. Glycoprotein IIb/IIIa inhibitors, bivalirudin and sodium nitroprusside will be administered at the discretion of the treating physician.

Measurements To analyze the ventricular dimensions, myocardium at risk (MaR) and infarct size, using postprocessing software, patients will be allocated to undergo cardiac magnetic resonance examinations at the core laboratory (the First Affiliated Hospital with Nanjing Medical University, Nanjing, China).

Troponin T/I, myoglobin, and creatine kinase-MB will be sampled before randomization and at 12 and 24 h after catheterization. We define the peak values as the highest measured values within 24 h by calculating under area of the curve from the measurements. N-terminal pro-brain natriuretic peptide will be sampled and dynamic electrocardiogram be performed at 48h after admission.

Clinical endpoints. Clinical events will be collected using a clinical report form during the index hospital stay, at 30±10 days, and at 12 months. Furthermore, adverse event and serious adverse event reporting will be collected as clinical endpoints. The independent monitors supervise hospital charts for all patients. All primary events (death, re-infarction, target lesion revascularization, major bleeding and heart failure) will be assessed independently by a blinded clinical events committee.

Statistical analysis. Calculations and statistics will be performed by using the GraphPad Prism 5.0 software (GraphPad Software Inc, La Jolla, Calif). The Fisher exact test will be performed on categorical variables. Continuous variables will be tested using Mann-Whitney Utest with exact inference. Statistical significance will be conducted at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients who present with an anterior or inferior STEMI with ST-segment elevation of 0.2 mV in >2 or more anatomically contiguous leads and a duration of symptoms of <6 hours are included.

-

Exclusion Criteria:

Participants with cardiac arrest, previous AMI, previous PCI or CABG, known congestive heart failure, end-stage kidney disease or hepatic failure, coagulopathy, pregnancy, or Killip class II through IV at presentation are excluded in this study.

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Infarct Size | The Infarct Size of Myocardial Is Measured by Magnetic Resonance Imaging in Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Lian-Sheng Wang, MD, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erlinge D, Gotberg M, Noc M, Lang I, Holzer M, Clemmensen P, Jensen U, Metzler B, James S, Botker HE, Omerovic E, Koul S, Engblom H, Carlsson M, Arheden H, Ostlund O, Wallentin L, Klos B, Harnek J, Olivecrona GK. Therapeutic hypothermia for the treatment of acute myocardial infarction-combined analysis of the RAPID MI-ICE and the CHILL-MI trials. Ther Hypothermia Temp Manag. 2015 Jun;5(2):77-84. doi: 10.1089/ther.2015.0009. Epub 2015 May 18. PMID 25985169
- [Background] Villablanca PA, Rao G, Briceno DF, Lombardo M, Ramakrishna H, Bortnick A, Garcia M, Menegus M, Sims D, Makkiya M, Mookadam F. Therapeutic hypothermia in ST elevation myocardial infarction: a systematic review and meta-analysis of randomised control trials. Heart. 2016 May;102(9):712-9. doi: 10.1136/heartjnl-2015-308559. Epub 2016 Feb 10. PMID 26864673
- [Background] Kohlhauer M, Berdeaux A, Ghaleh B, Tissier R. Therapeutic hypothermia to protect the heart against acute myocardial infarction. Arch Cardiovasc Dis. 2016 Dec;109(12):716-722. doi: 10.1016/j.acvd.2016.05.005. Epub 2016 Sep 28. PMID 27692660
- [Result] Kim H, Lee J, Song W, Shin J, Oh D, Harrison K, Jakkula M, Wong SC, Hong MK. Feasibility and safety of regional myocardial hypothermia during myocardial ischemia and infarction in pigs. Coron Artery Dis. 2005 Mar;16(2):125-9. doi: 10.1097/00019501-200503000-00008. PMID 15735406
- [Result] Otake H, Shite J, Paredes OL, Shinke T, Yoshikawa R, Tanino Y, Watanabe S, Ozawa T, Matsumoto D, Ogasawara D, Yokoyama M. Catheter-based transcoronary myocardial hypothermia attenuates arrhythmia and myocardial necrosis in pigs with acute myocardial infarction. J Am Coll Cardiol. 2007 Jan 16;49(2):250-60. doi: 10.1016/j.jacc.2006.06.080. Epub 2006 Dec 29. PMID 17222738
- [Result] Otterspoor LC, Van't Veer M, van Nunen LX, Wijnbergen I, Tonino PA, Pijls NH. Safety and feasibility of local myocardial hypothermia. Catheter Cardiovasc Interv. 2016 Apr;87(5):877-83. doi: 10.1002/ccd.26139. Epub 2015 Aug 13. PMID 26269225
- [Result] Erlinge D, Gotberg M, Lang I, Holzer M, Noc M, Clemmensen P, Jensen U, Metzler B, James S, Botker HE, Omerovic E, Engblom H, Carlsson M, Arheden H, Ostlund O, Wallentin L, Harnek J, Olivecrona GK. Rapid endovascular catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. The CHILL-MI trial: a randomized controlled study of the use of central venous catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. J Am Coll Cardiol. 2014 May 13;63(18):1857-65. doi: 10.1016/j.jacc.2013.12.027. Epub 2014 Feb 5. PMID 24509284
- [Result] Dixon SR, Whitbourn RJ, Dae MW, Grube E, Sherman W, Schaer GL, Jenkins JS, Baim DS, Gibbons RJ, Kuntz RE, Popma JJ, Nguyen TT, O'Neill WW. Induction of mild systemic hypothermia with endovascular cooling during primary percutaneous coronary intervention for acute myocardial infarction. J Am Coll Cardiol. 2002 Dec 4;40(11):1928-34. doi: 10.1016/s0735-1097(02)02567-6. PMID 12475451